CLINICAL TRIAL: NCT01909401
Title: Pilot Study With Peginterferon, Ribavirin, and Boceprevir Prior to Transplantation to Clear Virus in Hepatitis C Genotype 1 Infected Individuals Undergoing Orthotopic Liver Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1301010500
Record Dates: First submitted 2013-06-13; First posted 2013-07-26 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation
MeSH Terms: interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: boceprevir

SUMMARY:
Currently, there is no treatment standard for use of anti-HCV (hepatitic C virus) medications for those preparing for a liver transplant. The purpose of this study is to determine whether those individuals who require liver transplantation for Hepatitis C, genotype I, who are undergoing liver transplantation may successfully get rid of their virus before the transplant by taking three medicines, peginterferon, ribavirin, and boceprevir, up until the time of the liver transplant surgery. If successful, the Hepatitis C virus will not re-infect the new liver that they receive and they will not require therapy for Hepatitis C after liver transplantation. This study involves the use of peginterferon alfa-2b, ribavirin, and boceprevir, all of which are approved for the treatment of genotype I Hepatitis C.

Hypothesis: The addition of boceprevir to peginterferon alfa-2b and ribavirin in patients with Hepatitis C genotype 1 with or without hepatocellular carcinoma undergoing orthotopic liver transplantation will lead to rapid HCV RNA clearance of genotype I infected individuals. Transplantation with anhepatic boceprevir will prevent reinfection of the new transplanted graft and prevent graft infection posttransplantation.

DETAILED DESCRIPTION:
Subject Patient Inclusion Criteria: Men and women age 18 to 70 inclusive, patients with genotype I Hepatitis C who are listed for orthotopic liver transplantation (OLT) will be enrolled. Those with hepatocellular carcinoma with or without treatment of hepatoma may also be included. The MELD score for enrollment will be capped at 16. Patients must have medically controlled ascites and those who have moderate or poorly controlled ascites will be excluded.

Treatment Plan: Fifteen patients with chronic genotype I Hepatitis C will be enrolled. All patients will begin with peginterferon and ribavirin for 4 weeks with the addition of boceprevir after Week 4 until orthotopic liver transplantation. The dose of interferon will be peginterferon 1.0 mcg/kg with weight-based ribavirin (600-1200 mg) with boceprevir 800 mg TID (three times per day) until OLT. All patients will be listed for orthotopic liver transplantation. HCV RNA will be measured monthly. When they are called in for transplant, they will take their last dose of ribavirin just prior to going to operating room. Patients will undergo orthotopic liver transplantation under standard protocol by Indiana University. They will receive by Dobhoff boceprevir 800 tid for 3 doses post transplantation. Virologic failure will be HCV RNA > 100 I.U. at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-70
* Patients must be genotype I HCV-infected individuals with cirrhosis undergoing orthotopic liver transplantation.
* Those with hepatocellular carcinoma with or without treatment of hepatoma may also be included.
* The MELD score for enrollment will be capped at 16.
* Patients must have medically controlled ascites and those who have moderate or poorly controlled ascites will be excluded.

Inclusion Laboratory Values

ALT (alanine aminotransferase) < 250 IU/L, AST (Aspartate aminotransferase ) < 250 IU/L, total bilirubin < 3 mg/dl, creatinine clearance > 45 ml by MDRD (Modification of Diet in Renal Disease), albumin > 2.8 g/dl, hemoglobin > 11, white count > 2.0 X103, absolute neutrophil count 1.5 X103, platelet count > 50,000.

Women of childbearing potential and male patients with sexual female partner who is of childbearing potential should use two acceptable methods of contraception.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of individuals who can remain HCV RNA undetected 6 months post orthotopic liver transplant after receiving peginterferon, ribavirin, and boceprevir. | 6 months post orthotopic liver transplant
  The primary objective is to determine the number of individuals who can remain HCV RNA undetected 6 months post orthotopic liver transplant after receiving peginterferon, ribavirin, and boceprevir. The primary safety objective is to determine the safety and efficacy of peginterferon, ribavirin, and boceprevir in Hepatitis C, genotype I individuals undergoing orthotopic liver transplantation.

SECONDARY OUTCOMES:
Safety and efficacy of peginterferon, ribavirin, and boceprevir in patients with genotype I undergoing orthotopic liver transplant for cirrhosis and/or hepatocellular carcinoma. | 6 months post orthotopic liver transplant
  To determine the safety and efficacy of peginterferon, ribavirin, and boceprevir in patients with genotype I undergoing orthotopic liver transplant for cirrhosis and/or hepatocellular carcinoma as defined by incidence of severe infections (SBP, bacteremia) and new onset ascites and or encephalopahty.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Kwo, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine - IUHealth-University Hospital, Indianapolis, Indiana, United States